CLINICAL TRIAL: NCT00667849
Title: Trial to Evaluate UltraSound in the Treatment of Tibial Fractures
Acronym: TRUST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to futility
Sponsor: Bioventus LLC (Industry)
Collaborators: McMaster University (Other); Clinical Advances Through Research and Information Translation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX-TIB-0907
Record Dates: First submitted 2008-04-21; First posted 2008-04-28 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Tibial Fractures
Keywords: Tibia
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exogen 4000+ (Active Comparator): Single arm, Exogen 4000+
  Interventions: Device: Exogen 4000+
- Sham (Sham Comparator): Single arm, sham (identical device with the exception of administration of ultrasound).
  Interventions: Device: Sham

INTERVENTIONS:
Device: Exogen 4000+ — Low-intensity pulsed ultrasound (LIPUS)
  Other Names: Exogen Bone Healing System - 4000+ series
  Arms: Exogen 4000+
Device: Sham — sham device identical to active device with the exception of administration of ultrasound
  Other Names: Single arm, sham of the Exogen 4000+
  Arms: Sham

SUMMARY:
The purpose of this study is to determine the effect of low-intensity, pulsed ultrasound on tibial fractures treated with intramedullary nailing.

DETAILED DESCRIPTION:
A randomized, placebo controlled, clinical trial to evaluate the safety and efficacy of low-intensity, pulsed ultrasound, applied to tibial fractures treated with intramedullary nailing.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 years or older
* Have an open or closed tibial fracture amenable to intramedullary nail fixation

Exclusion Criteria:

* Tibial fracture associated with a vascular injury requiring repair
* Pilon fractures
* Tibial fractures that extend into the joint and require reduction
* Pathologic fractures • Bilateral tibial fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, Principal Investigator — McMaster University
Locations (16):
- United States (13):
  - San Francisco General/Dept of Orthopedic Surgery, San Francisco, California
  - Florida Orthopedic Institute, Tampa, Florida
  - OrthoIndy, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Missouri, Columbia, Missouri
  - Insall Scott Kelly Institute, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rothman Institute, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Orthopedic Specialtiy Associates, Fort Worth, Texas
  - West Virginia University, Morgantown, West Virginia
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver Coastal Health, Vancouver, British Columbia
  - QE II Health Sciences Centre, Halifax, Nova Scotia

REFERENCES:
- [Derived] Findakli F, Busse JW, Schemitsch EH, Lonn E, Farrokhyar F, Bhandari M; and the TRUST Investigators. Smoking, Obesity, and Disability Benefits or Litigation Are Not Associated with Clinically Important Reductions in Physical Functioning After Intramedullary Nailing of Tibial Shaft Fractures: A Retrospective Cohort Study. Clin Orthop Relat Res. 2021 Apr 1;479(4):805-813. doi: 10.1097/CORR.0000000000001573. PMID 33196584
- [Derived] TRUST Investigators writing group; Busse JW, Bhandari M, Einhorn TA, Schemitsch E, Heckman JD, Tornetta P 3rd, Leung KS, Heels-Ansdell D, Makosso-Kallyth S, Della Rocca GJ, Jones CB, Guyatt GH. Re-evaluation of low intensity pulsed ultrasound in treatment of tibial fractures (TRUST): randomized clinical trial. BMJ. 2016 Oct 25;355:i5351. doi: 10.1136/bmj.i5351. PMID 27797787
- [Derived] Busse JW, Bhandari M, Einhorn TA, Heckman JD, Leung KS, Schemitsch E, Tornetta P 3rd, Walter SD, Guyatt GH. Trial to re-evaluate ultrasound in the treatment of tibial fractures (TRUST): a multicenter randomized pilot study. Trials. 2014 Jun 4;15:206. doi: 10.1186/1745-6215-15-206. PMID 24898987
- [Derived] Dijkman BG, Busse JW, Walter SD, Bhandari M; TRUST Investigators. The impact of clinical data on the evaluation of tibial fracture healing. Trials. 2011 Nov 3;12:237. doi: 10.1186/1745-6215-12-237. PMID 22050862

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham: Single arm, sham (identical to active device with the exception of administration of ultrasound)
  Sham: sham device identical to active device with the exception of administration of ultrasound
Period: Overall Study
Arm/Group | Exogen 4000+ | Sham
Started | 250 | 251
Completed | 142 | 130
Not Completed | 108 | 121

BASELINE CHARACTERISTICS:
Groups:
- Sham: Single arm, sham (identical to active device with the exception of administration of ultrasound).
  Sham: sham device identical to active device with the exception of administration of ultrasound
- Total: Total of all reporting groups
Arm/Group | Exogen 4000+ | Sham | Total
Number analyzed (Participants) | 250 | 251 | 501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 244 | 239 | 483
  >=65 years | 6 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (13.2) | 39.1 (14.6) | 38.3 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 75 | 156
  Male | 169 | 176 | 345
Region of Enrollment [Number; unit: participants]
  Canada | 82 | 85 | 167
  United States | 168 | 166 | 334

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the SF-36 Physical Component Summary (PCS) Score of the Short Form-36 (SF-36)
Description: Assessments at baseline and 6 post baseline time points/ mixed effects repeated measure single point estimate. Range= -100 worst, 0 best
Time Frame: Over 365 days
Population: Full Analysis Set (FAS) is all subjects randomized with at least one post treatment set of adjudicated x-rays.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Exogen 4000+: Single arm, active Exogen 4000+ Low-intensity pulsed ultrasound (LIPUS)
- Sham: Single arm, sham (identical to active device with the exception of administration of ultrasound)
Arm/Group | Exogen 4000+ | Sham
Number analyzed (Participants) | 241 | 242
units on a scale | -6.9 [-8.0 to -5.9] | -7.5 [-8.6 to -6.5]

2. Primary Outcome: Time (Days) to Radiographic Healing of Tibial Fractures
Description: Days from randomization to day of x-ray assessed healed or, if not healed, day of premature withdrawal/study termination or day 365 (end of study visit)/ Kaplan-Meier
Time Frame: over 365 days
Population: Full Analysis Set (FAS) is all subjects randomized with at least one post treatment set of adjudicated x-rays.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Sham: Single arm, sham (identical to active device with the exception of administration of ultrasound)
  Sham: device identical to active device with the exception of administration of ultrasound
Arm/Group | Exogen 4000+ | Sham
Number analyzed (Participants) | 241 | 242
days | 130 [112 to 183] | 133 [115 to 186]

3. Other Pre Specified Outcome: Treatment Compliance
Description: The percent of subjects who used the device greater than or equal to 18 minutes per day over 80% of the days in their treatment period.
Time Frame: Treatment period: Days from randomization to day of x-ray assessed healed or, if not heal, day of premature withdrawal/study termination or day 365 (end of study visit)
Population: FAS with compliance data (subjects who returned the device)
Measure: Number; unit: percentage of compliant participants
Arm/Group | Exogen 4000+ | Sham
Number analyzed (Participants) | 213 | 215
percentage of compliant participants | 44.6 | 42.3

ADVERSE EVENTS:
Time Frame: up to 2 years
Description: no standardized coding dictionary used
Groups:
- Exogen 4000+: Single arm, active Exogen 4000+ ultrasound bone healing system
  Low-intensity pulsed ultrasound (LIPUS)
Arm/Group | Exogen 4000+ | Sham
Serious Adverse Events (participants affected / at risk) | 3/250 | 5/251
Other Adverse Events (participants affected / at risk) | 98/250 | 97/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exogen 4000+ (N=250) | Sham (N=251)
acute chest pain (Cardiac disorders) | 0 (0) | 1 (1) — abnormal troponin level and nausea Resulted in hospitalization Not related to device
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) — Resulted in hospitalization Not related to device
Infection, tissue (Infections and infestations) | 1 (1) | 0 (0) — Resulted in hospitalization, was a life threatening situation, necessitated medical surgical intervention to preclude primary impairment of body function or permanent damage to a body structure. Not related to device.
Renal dysfunction (creatinine 2x BL level (Renal and urinary disorders) | 0 (0) | 1 (1) — Resulted in hospitalization Not related to device
Broken screw (Surgical and medical procedures) | 1 (1) | 1 (1) — Resulted in hospitalization Not related to device
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — tendonitis of hip; resulted in hospitalization
sternal wire closure disruption (Cardiac disorders) | 0 (0) | 1 (1) — resulted in hospitalization
cough, vomiting, leukocytosis, increased troponin (Gastrointestinal disorders) | 0 (0) | 1 (1) — possible gastroenteritis resulted in hospitalization
infection tissue (Infections and infestations) | 0 (0) | 1 (1) — cellulitis; resulted in hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exogen 4000+ (N=250) | Sham (N=251)
Edema (Blood and lymphatic system disorders) | 18 (18) | 15 (16) — Edema of left lower extremity
Other, not listed on AE form (General disorders) | 7 (7) | 21 (24)
Pain (General disorders) | 8 (8) | 8 (8)
Infection, tissue (Infections and infestations) | 6 (6) | 9 (9)
Wound complication (Infections and infestations) | 7 (7) | 5 (5)
accident/fall (Injury, poisoning and procedural complications) | 14 (15) | 7 (7)
Non-union (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (5)
Other local event (Musculoskeletal and connective tissue disorders) | 19 (19) | 20 (21)
Pain (Nervous system disorders) | 48 (58) | 49 (63)
Rash/redness at treated area (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)

LIMITATIONS AND CAVEATS:
Poor Compliance: Protocol defined compliance as ≥18 minutes use per day. Devices have a treatment monitor that showed average compliance of 42.3% (sham) and 44.6% (active) in 80% of treatment days. Poor treatment adherence confounds results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less